CLINICAL TRIAL: NCT00759200
Title: An Open-label, Randomized, Multicenter, Active-controlled, Dose-ranging Study to Evaluate the Safety and Efficacy of Albinterferon Alfa 2b Administered Every 4 Weeks Plus Ribavirin in Interferon Alfa-naïve Patients With Genotype 2/3 Chronic Hepatitis C
Brief Title: Safety and Efficacy of Albumin Interferon Administered Every 4 Weeks in Genotype 2/3 Hepatitis C Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABF656B2202
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; genotype 2; genotype 3; albumin interferon alfa-2b; alb-interferon
MeSH Terms: conditions — Hepatitis C, Chronic

ARMS (5):
- alb-interferon arm 1 (Experimental)
  Interventions: Drug: alb-interferon alfa 2b
- alb-interferon arm 2 (Experimental)
  Interventions: Drug: alb-interferon alfa 2b
- alb-interferon arm 3 (Experimental)
  Interventions: Drug: alb-interferon alfa 2b
- alb-interferon arm 4 (Experimental)
  Interventions: Drug: alb-interferon alfa 2b
- peg-interferon (Active Comparator)
  Interventions: Drug: peg-interferon

INTERVENTIONS:
Drug: alb-interferon alfa 2b — 900 mcg every 4 weeks
  Other Names: ABF656
  Arms: alb-interferon arm 1
Drug: alb-interferon alfa 2b — 1200 mcg every 4 weeks
  Other Names: ABF656
  Arms: alb-interferon arm 2
Drug: alb-interferon alfa 2b — 1500 mcg every 4 weeks
  Other Names: ABF656
  Arms: alb-interferon arm 3
Drug: alb-interferon alfa 2b — 1800 mcg every 4 weeks
  Other Names: ABF656
  Arms: alb-interferon arm 4
Drug: peg-interferon — Peg-interferon alfa 2a: 180 mcg 1x per wk.
  Other Names: peg-IFN
  Arms: peg-interferon

SUMMARY:
This study will evaluate the safety and efficacy of alb-interferon in adults with genotype 2 or 3 chronic hepatitis

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Clinical diagnosis of chronic hepatitis C
* Infection with HCV genotype 2 or 3
* No previous IFNα-based therapy

Exclusion Criteria:

* Women of child-bearing potential if not using double barrier method of contraception, pregnant or nursing
* Fertile males, unless condom with spermicide is used and female partner agrees to use one or more of the acceptable methods until 7 months after last dose of RBV
* History or current evidence of decompensated liver disease; other forms of liver disease
* Coinfection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* History of moderate, severe or uncontrolled psychiatric disease
* History of seizure disorder
* History or clinical evidence of chronic cardiac disease, preexisting interstitial lung disease or severe lung disease
* Clinically significant findings on eye/retinal examination
* History of immunologically mediated disease
* Organ transplantation other than cornea or hair transplant
* History of clinically significant hemoglobinopathy
* Diagnosis of malignancy of any organ system with the exception of localized basal cell carcinoma of the skin
* History of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* Drug or alcohol addiction within the last 6 months and/or positive drug screening tests
* Received systemic corticosteroids (prednisone equivalent of > 10 mg/day) within 14 days prior to Baseline visit
* Received concomitant systemic antibiotics, antifungals or antivirals for the treatment of active infection within 14 days prior to Baseline visit.
* Received herbal therapies (including milk thistle or glycyrrhizin) or an investigational drug within 35 days prior to Baseline visit
* Have a clinically significant laboratory abnormality

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | at every visit

SECONDARY OUTCOMES:
Viral load | at weeks 4, 12 and 24 of treatment and 24 weeks post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- Australia (6):
  - Novartis Investigative site, Clayton
  - Novartis Investigative site, Fitzroy
  - Novartis Investigative site, Greenslopes
  - Novartis Investigative site, Kingswood
  - Novartis Investigative site, Melbourne
  - Novartis Investigative site, Westmead
- Canada (5):
  - Novartis Investigative site, Calgary
  - Novartis Investigative Site, Downsview
  - Novartis Investigative site, Montreal
  - Novartis Investigative site, Toronto
  - Novartis Investigative site, Vancouver
- France (4):
  - Novartis Investigative Site, Cretail
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
- Greece (5):
  - Novartis Investigative Site, Heraklion
  - Novartis Investigative Site, Loannina
  - Novartis Investigative Site, Patra-Rio
  - Novartis Investigative Site, Piraeurs
  - Novartis Investigative Site, Thessaloniki
- India (6):
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative site, Hyderabad
  - Novartis Investigative Site, Lucknow
  - Novartis Investigative Site, Ludhiana
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
- Italy (7):
  - Novartis Investigative site, Bologna
  - Novartis Investigative site, Milan
  - Novartis Investigative site, Napoli
  - Novartis Investigative site, Pavia
  - Novartis Investigative site, Pisa
  - Novartis Investigative site, Polermo
  - Novartis Investigative site, Torino
- Poland (2):
  - Novartis Investigative site, Bialystok
  - Novartis Investigative site, Lodz
- Spain (6):
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Madrid
  - Novartis Investigative site, Málaga
  - Novartis Investigative site, Oviedo
  - Novartis Investigative site, Seville
  - Novartis Investigative site, Valencia
- Taiwan (3):
  - Novartis Investigative site, Kaohsiung City
  - Novartis Investigative site, Tainan
  - Novartis Investigative site, Taipei
- Thailand (4):
  - Novartis Investigative site, Bangkok
  - Novartis Investigative site, Chaingmai
  - Novartis Investigative Site, Hat Yai
  - Novartis Investigative Site, Muang
- Novartis Investigative Site, Glasgow, United Kingdom

REFERENCES:
- [Result] Pianko S, Zeuzem S, Chuang WL, Foster GR, Sarin SK, Flisiak R, Lee CM, Andreone P, Piratvisuth T, Shah S, Sood A, George J, Gould M, Komolmit P, Thongsawat S, Tanwandee T, Rasenack J, Li Y, Pang M, Yin Y, Feutren G, Jacobson IM; B2202 Study Team. Randomized trial of albinterferon alfa-2b every 4 weeks for chronic hepatitis C virus genotype 2/3. J Viral Hepat. 2012 Sep;19(9):623-34. doi: 10.1111/j.1365-2893.2012.01586.x. Epub 2012 Mar 21. PMID 22863266